CLINICAL TRIAL: NCT01353144
Title: A Comparison of Two Therapeutic Strategies for the Treatment of Aspirin-associated Peptic Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS96-CT4-26
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Results first posted 2015-10-14 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-09

CONDITIONS: Peptic Ulcer
Keywords: aspirin; peptic ulcer
MeSH Terms: conditions — Peptic Ulcer | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- esomeprazole (No Intervention): esomeprazole (40 mg/day) for 8 weeks
- esomeprazole plus aspirin (Active Comparator): esomeprazole (40 mg/day) plus aspirin (100 mg/day) for 8 weeks
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin — aspirin, 100 mg, qd x 8 weeks
  Other Names: aspirin protect
  Arms: esomeprazole plus aspirin

SUMMARY:
Esomeprazole plus aspirin compared with esomeprazole alone for the treatment of aspirin-related peptic ulcers.

DETAILED DESCRIPTION:
The aims of this study are to compare esomeprazole plus aspirin with esomeprazole alone in the treatment of aspirin-related ulcers.

Patients with aspirin-related peptic ulcers are randomized to receive esomeprazole (40 mg/day) plus aspirin (100 mg/day) or esomeprazole (40 mg/day) alone for 8 weeks. Follow-up endoscopy was carried out at the end of the eighth week. The primary end point was the healing of peptic ulcers.

ELIGIBILITY:
Inclusion Criteria:

* aspirin users who have a peptic ulcer confirmed by endoscopy

Exclusion Criteria:

* serious medical illness (including cardiovascular events within 6 months before endoscopy)
* acute gastrointestinal bleeding
* a history of gastric or duodenal surgery
* allergic to the study drugs
* require long-term treatment with non-aspirin nonsteroidal anti-inflammatory drugs (NSAIDs), antiplatelet agents, or anticoagulant agents
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwok-Hung Lai, MD, Study Chair — Kaohsiung Veterans General Hospital.
Locations (3):
- Taiwan (3):
  - Chung-Ho Hospital, Kaohsiung, Taiwan
  - Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan
  - Kaohsiung Veterans General Hospital, Kaohsiung City

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Esomeprazole | Esomeprazole Plus Aspirin
Started | 89 | 89
Completed | 80 | 81
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Esomeprazole Plus Aspirin | Total
Number analyzed (Participants) | 89 | 89 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 26 | 47
  >=65 years | 68 | 63 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (11.0) | 69.9 (12.4) | 69.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 53 | 52 | 105
Region of Enrollment [Number; unit: participants]
  Taiwan | 89 | 89 | 178

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Whom Peptic Ulcer Was Healed
Description: Number of participants in whom peptic ulcer was healed at week 8
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Esomeprazole Plus Aspirin
Number analyzed (Participants) | 89 | 89
participants | 66 | 66

2. Secondary Outcome: Number of Participants Deveoping Peptic Ulcer Bleeding
Description: Number of participants deveoping peptic ulcer bleeding during 8-week study period
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Esomeprazole Plus Aspirin | Esomeprazole
Number analyzed (Participants) | 89 | 89
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Esomeprazole | Esomeprazole Plus Aspirin
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 1/89 | 2/89
OTHER ADVERSE EVENTS (reported when occurring in more than 1.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esomeprazole (N=89) | Esomeprazole Plus Aspirin (N=89)
skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
persistent dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes